CLINICAL TRIAL: NCT01255943
Title: Testing Spread and Implementation of Novel MRSA-Reducing Practices
Brief Title: Testing Spread and Implementation of Novel Methicillin Resistant Staphylococcal Aureus (MRSA)-Reducing Practices
Status: Completed | Type: Observational
Sponsor: MaineHealth (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Mark Parker, Director, Division of Nephrology and Transplantation, MaineHealth
Other Study IDs: HHSA290200600013
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Blood Stream Infections; MRSA Infections
Keywords: MRSA; bloodstream infections; hemodialysis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- prevalent hemodialysis patients: These patients are observed in two outpatient dialysis units with a combined census of approximately 175 patients
  Interventions: Behavioral: healthcare staff processes for infection prevention

INTERVENTIONS:
Behavioral: healthcare staff processes for infection prevention — Toyota lean and positive deviance discovery and action dialogues to facilitate process improvement

SUMMARY:
The purpose of this study is to implement strategies for improved efficiency and waste reduction ("Toyota Lean") and positive deviance, a social behavioral change process, utilizing frontline healthcare personnel to reduce infection bloodstream infection and MRSA infection in outpatient dialysis care. In two outpatient dialysis units, dialysis unit healthcare staff will be educated in Toyota lean techniques and conduct periodic "discovery and action" dialogues to identify and implement care process changes to reduce infection. Outcomes to be monitored will include incidence of bloodstream infections and MRSA infections of all types. Data will be assessed at quarterly intervals using interrupted time series analysis.

ELIGIBILITY:
Inclusion Criteria: all hemodialysis patients at two outpatient dialysis units

Exclusion Criteria:peritoneal dialysis patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: prevalent hemodialysis patients at two outpatient dialysis units
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of bloodstream infections | 14 months

SECONDARY OUTCOMES:
Incidence of MRSA infections | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Parker, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States